CLINICAL TRIAL: NCT00972088
Title: Prevalence of Inflammatory Bowel Disease in Patients With Perianal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bikkur Holim Hospital (Other)
Responsible Party: Principal Investigator, Sam Adler, Prof. Samuel N. Adler, MD, Bikkur Holim Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Peri Anal Study
Record Dates: First submitted 2009-09-02; First posted 2009-09-04 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-05

CONDITIONS: Inflammatory Bowel Disease; Perianal Fistula; Perianal Abscess
Keywords: inflammation of the small bowel
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Capsule Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- capsule endoscopy (Other): patients eligible according to inclusion criteria who underwent a capsule endoscopy
  Interventions: Device: capsule endoscopy

INTERVENTIONS:
Device: capsule endoscopy — The disposable, ingestible PillCam® SB2 Capsule acquires the video images during natural propulsion through the digestive system. The Capsule transmits the acquired images via digital radio frequency communication channel to the Given® Data Recorder unit located outside the body.

SUMMARY:
To show that prevalence of inflammation of the small bowel in patients with anorectal disease is under-diagnosed based on colonoscopy ileoscopy alone.

DETAILED DESCRIPTION:
IBD of the small bowel is associated with perianal disease such as ano-rectal abscesses and fistulas. Colonoscopy with ileoscopy and small bowel series are relied upon to document the presence of Crohn's disease of the small bowel. We suspect that the prevalence of inflammatory small bowel disease is underestimated.

In my practice I have cases that had negative colonoscopy ileoscopy and positive findings at capsule endoscopy. These patients are receiving therapy for Crohn's disease. It is important to prove that the prevalence is higher.

Capsule Endoscopy (CE) is the "first line tool" diagnostic procedure for the examination of the small bowel. It is performed today in more than 2,900 GI clinics in hospitals, outpatient departments and physicians' offices all over the world using the PillCam® Platform. Over 500,000 CE procedures with the Given PillCam SB have been completed to date.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 10 - 80
* Patients with anorectal abscess of anorectal fistula
* Patient is male or female
* Within three months prior to enrollment, patient has normal test results for at least one of the following tests:

  1. Colonoscopy with Ileoscopy, and/or
  2. Colonoscopy with small bowel series, and/or
  3. Colonoscopy with CT enterography
* Within three months prior to enrollment patient has the following lab tests: Blood count, sedimentation rate, CRP. IBD serology is optional.
* Sign informed consent

Exclusion Criteria:

* Can not sign informed consent
* Contraindications to colonoscopy ileoscopy or capsule endoscopy
* History of established IBD

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Adler, Prof., Principal Investigator — Bikur Cholim Hospital, Jerusalem
Locations (3):
- Israel (3):
  - Assaf Harofeh Medical Center, Tel Aviv, Zrifin
  - Rambam Medical Center, Haifa
  - Bikur Cholim Hospital, Jerusalem

RESULTS

PARTICIPANT FLOW:
Recruitment Details: from 2009 until june 2011 26 patients were enrolled from gastroenterology clinics
Pre-assignment Details: patients were enrolled to undergo capsule endoscopy of the small bowel if they had perianal disease and a negative colonoscopy with ileoscopy or a negative colonoscopy with a negative small bowel series or negative ct enterography
Groups:
- a Single Arm Group, Patients With Ano Rectal Disease: patients suffering from anorectal disease with a negative standard work up to rule out crohn's disease
Period: Overall Study
Arm/Group | a Single Arm Group, Patients With Ano Rectal Disease
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Anorectal Disease, Negative Work up for Crohns Disease: Patients presently suffering from anorectal abscess or anorectal fistula
Arm/Group | Anorectal Disease, Negative Work up for Crohns Disease
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 34.3 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 17
Region of Enrollment [Number; unit: participants]
  Israel | 26

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Inflammation as Diagnosed by Capsule Endoscopy
Description: The capsule endoscopy findings were carefully examined by specialists in the field. findings such as erosions, edema, erythema and ulceration in significant areas of the intestine led to the clinical diagnosis of crohn's disease. all together 6 patients were diagnosed as suffering from crohn's disease.
Time Frame: up to 7 days
Population: per protocol
Measure: Number; unit: participants
Arm/Group | Anorectal Disease, Negative Work up for Crohns Disease
Number analyzed (Participants) | 26
participants | 6

ADVERSE EVENTS:
Arm/Group | Anorectal Disease, Negative Work up for Crohns Disease
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes